CLINICAL TRIAL: NCT01536314
Title: Preventing the Development of Neuropathic Pain Post-mastectomy/Tumorectomy by Pre-emptive or Post-operative Memantine Administration
Brief Title: Prophylaxis of Neuropathic Pain by mémantine
Acronym: MEMANTINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0115
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Neuropathic Pain
Keywords: Pre-emptive administration; Post-operative administration; Prophylaxis; Memantine; Post-mastectomy/tumorectomy; Neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Memantine

INTERVENTIONS:
Drug: Memantine EBIXA® — The aim of this study is to evaluate if memantine administered during 4 weeks beginning 2 weeks before surgery induces a decrease of painful intensity 3 months after surgery, compared to placebo group.
Drug: Placebo : lactose — The aim of this study is to evaluate if memantine administered during 4 weeks beginning 2 weeks before surgery induces a decrease of painful intensity 3 months after surgery, compared to placebo group.

SUMMARY:
The aim of this study is to evaluate if memantine administered during 4 weeks beginning 2 weeks before surgery induces a decrease of painful intensity 3 months after surgery, compared to placebo group.

DETAILED DESCRIPTION:
The aim of this study is to evaluate if memantine administered during 4 weeks beginning 2 weeks before surgery induces a decrease of painful intensity 3 months after surgery, compared to placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* patient suffering breast cancer with mastectomy/tumorectomy with or within cleaning 2 weeks after inclusion with or within pre-emptive chemotherapy

Exclusion Criteria:

* Against-indication at memantine administration : hypersensitivity at active substance or excipients, hypertension, antecedent cerebrovascular accident, severe cardiac insufficiency
* Diabetic patient (Type I and II)
* Patient with medical or surgical antecedents
* Patient receiving treatment with amantadine, ketamine, dextrometorphan, L-Dopa, dopaminergic, anticholinergic agonists, barbiturate, neuroleptic, IMAO, antispastic agents, dantrolen or baclofen, phenitoin, cimetidine, ranitidine, procainamide, quinidine, quinine, nicotine, hydrochlorothiazide, warfarine
* Patient with alcohol addiction
* Woman in childbearing age not using effective contraceptive method, pregnant or lactating woman
* Patient who participated in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
average painful intensity | 5 days before visit of 3 months

SECONDARY OUTCOMES:
Evaluation of pain by numerical scale | during 15 first days following surgery and to visit of 3 months
Average painful | on 5 days before visit of 6 months post-surgery
analgesic consumption | during 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Morel V, Joly D, Villatte C, Dubray C, Durando X, Daulhac L, Coudert C, Roux D, Pereira B, Pickering G. Memantine before Mastectomy Prevents Post-Surgery Pain: A Randomized, Blinded Clinical Trial in Surgical Patients. PLoS One. 2016 Apr 6;11(4):e0152741. doi: 10.1371/journal.pone.0152741. eCollection 2016. PMID 27050431
- [Derived] Pickering G, Morel V, Joly D, Villatte C, Roux D, Dubray C, Pereira B. Prevention of post-mastectomy neuropathic pain with memantine: study protocol for a randomized controlled trial. Trials. 2014 Aug 20;15:331. doi: 10.1186/1745-6215-15-331. PMID 25142039